CLINICAL TRIAL: NCT03776539
Title: A Phase 1, Open-label, Single-dose, Parallel-group Study to Evaluate the Effects of Renal Impairment on the Pharmacokinetics of ELX-02
Brief Title: A Study to Evaluate the Effects of Renal Impairment on the Pharmacokinetics of ELX-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eloxx Pharmaceuticals, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EL-008
Record Dates: First submitted 2018-12-04; First posted 2018-12-14 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Impaired Renal Function
Keywords: Impaired Renal Function; PK
MeSH Terms: conditions — Renal Insufficiency | interventions — ELX-02

STUDY DESIGN:
Intervention Model Description: Subjects will be categorized in 4 groups:
  Group 1: subjects with mild renal impairment
  Group 2: subjects with moderate renal impairment
  Group 3: subjects with severe renal impairment
  Group 4 (control group): subjects with normal renal function
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX-02 (Experimental): Drug: ELX-02
  Interventions: Drug: ELX-02

INTERVENTIONS:
Drug: ELX-02 — ELX-02 is a synthetic, designer eukaryotic ribosomal specific glycoside (ERSG) optimized as a translational read-through drug. All groups will get the same treatment.

SUMMARY:
Phase 1 - Pharmacokinetics in Patients with Impaired Renal Function

DETAILED DESCRIPTION:
The study is a two-center, Phase 1, open-label, single-dose, one-period, four-parallel-group, PK study in subjects with various severities of renal dysfunction and healthy volunteers.

Subjects will be categorized in 4 groups:

Group 1: subjects with mild renal impairment Group 2: subjects with moderate renal impairment Group 3: subjects with severe renal impairment Group 4 (control group): subjects with normal renal function

The mild (group 1) and moderate (group 2) patients with renal disease will be dosed first, in a parallel fashion. At this point, interim PK analyses will be performed and a safety committee composed of Sponsor and Contract Research Organization (CRO) members will jointly review the PK data before dosing the patients with severe renal disease (group 3). Control subjects (group 4) will be recruited after the recruitment of groups 1 to 3.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker and/or light smoker
2. Have a diagnosis of renal impairment that has been stable, without any significant change in overall disease status in the last 3 months prior to screening.
3. Have an estimated glomerular filtration rate (eGFR) expressed in mL/min/1.73 m2 (Modification of Diet in Renal Disease 4-variable [MDRD4] equation) at screening within the range of:

   1. Group 1 - Mild Group: 60 - 89 mL/min/1.73 m2;
   2. Group 2 - Moderate Group: 30 - 59 mL/min/1.73 m2;
   3. Group 3 - Severe Group: < 30 mL/min/1.73 m2 not requiring dialysis. eGFR results that are deemed inconsistent with the usual stage of renal impairment may be repeated. Subjects are categorized into severity group at screening. If the eGFR scores change on Day-1 or other visit due to a non-clinically significant change in clinical status or laboratory result, the subject keeps the original severity group.
4. Subject may have stable treated medical illnesses and underlying diseases producing the renal impairment such as diabetes, hypertension, or cardiovascular disease, providing that, in the opinion of the PI, the disease is stable.
5. Have normal or non-clinically significant findings at physical examination, vital signs and electrocardiogram (ECG) and normal limits or non-clinically significant deviations in clinical laboratory evaluations at screening.
6. Other than renal impairment, have no other conditions which may significantly impact study drug absorption or metabolism.
7. Stable medical regimen, deemed not to interact with study drug PK, for 14 days prior to dosing, except for routine daily management of electrolytes (e.g. potassium), acid-base, or other associated disorders expected in patients with renal impairment.
8. Females of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized since at least 6 months) must be willing to use acceptable contraceptive method throughout the study and for 30 days after study drug administration.
9. Male subjects who are not vasectomized for at least 6 months, and who are sexually active with a non-sterile female partner (sterile female partners include post-menopausal females and surgically sterile females) must be willing to use acceptable contraceptive method from dosing until at least 90 days after study drug administration.
10. Male subjects (including men who have had vasectomy) with a pregnant partner must agree to use a condom from dosing until at least 90 days after study drug administration.
11. Male subjects must be willing not to donate sperm until 90 days following study drug administration.
12. Able to understand and willing to sign the Informed Consent Form (ICF) and comply with the study restrictions.

Exclusion Criteria:

1. Unstable renal function or acute exacerbation of renal disease within 14 days of study drug administration, as indicated by recent history or worsening of clinical and/or laboratory signs of renal impairment.
2. Has a functioning renal transplant.
3. Major illness or surgery within 4 weeks prior to dosing.
4. Clinically significant unstable medical condition or history of any illness that may increase the risk associated with study participation or investigational drug administration or may interfere with the interpretation of study results and would make the subject inappropriate for entry into this study.
5. Positive test for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) at screening.
6. History of allergic reactions, hypersensitivity or toxic reactions to aminoglycosides.
7. History of anaphylaxis.
8. Supine 12-lead ECG abnormalities at screening considered clinically significant.
9. Clinically significant vital sign abnormalities at screening.
10. History of significant drug or alcohol abuse within six months prior to screening.
11. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days (or 5 half-lives, whichever is longer) prior to dosing, administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
12. Positive urine drug screen or alcohol test at screening.
13. Female subject with positive pregnancy test at screening.
14. Breast-feeding or pregnant subject within 6 months prior to study drug administration.
15. Use of any drugs known as strong inducer or inhibitor of hepatic drug metabolism within 30 days prior to study drug administration.
16. Use of medication other than stable medications approved by the PI and topical products without significant systemic absorption.
17. Use of prohibited medications as directed in the protocol.
18. Donation of plasma within 7 days prior to dosing. Donation or loss of blood within 30 days prior to the first dosing.
19. Any reason which, in the opinion of the PI, would prevent the subject from participating in the study.
20. Inability to be venipunctured and/or tolerate catheter venous access.
21. Presence of mitochondrial mutation(s) making the subject susceptible to aminoglycoside toxicity.
22. Presence of signs of dehydration, recent history of neuromuscular blockade or clinically significant history of vestibular impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Inventiv Health Clinical -Research Pharmacy Unit, Miami, Florida
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Eloxx Pharmaceuticals Website — http://www.eloxxpharma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were treated at medical clinics. Groups 1-2 Screening start: January 4, 2019 Screening end: 8 April 2019 Group 3 Screening start: 9 May 2019 Screening end: 17 June 2019 Group 4 Screening start: 26 June 2019 Screening end: 30 June 2019
Groups:
- Mild Renal Impairment: eGFR 60 to 89 mL/min/1.73 m^2
- Moderate Renal Impairment: eGFR 30 to 59 mL/min/1.73 m^2
- Severe Renal Impairment: eGFR <30 mL/min/1.73 m^2, Not Requiring Dialysis
- Healthy Volunteers: eGFR >=90 mL/min/1.73 m^2
Period: Overall Study
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Healthy Volunteers
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Mild Renal Impairment eGFR 60 to 89 mL/min/1.73 m^2
- Group 2: Moderate Renal Impairment eGFR 30 to 59 mL/min/1.73 m^2
- Group 3: Severe Renal Impairment eGFR <30 mL/min/1.73 m^2, Not Requiring Dialysis
- Group 4: Healthy Volunteers eGFR >=90 mL/min/1.73 m^2
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (5.9) | 65.0 (10.4) | 61.8 (8.2) | 57.7 (2.1) | 62.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 2 | 8
  Male | 4 | 3 | 5 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 6 | 5 | 22
  Not Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24
eGFR [Mean (Standard Deviation); unit: mL/min/1.73 m2] | 74.72 (9.25) | 40.07 (4.54) | 16.92 (9.77) | 100.25 (15.65) | 57.99 (34.06)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameters- Plasma AUC0-24
Description: Area under the curve (AUC0-24) of ELX-02 plasma concentration following a single subcutaneous (SC) dose
Time Frame: 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, and 24 hours after dosing
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*h/mL | 16877.94 (1714.57) | 32787.41 (7410.46) | 64895.29 (16967.68) | 15506.68 (3444.66)

2. Primary Outcome: Pharmacokinetic Parameters- Plasma Cmax
Description: Peak Plasma Concentration (Cmax) of ELX-02 following a single subcutaneous (SC) dose in subjects with normal renal function, mild, moderate, or severe renal impairment
Time Frame: 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24, 36, 48, 72, and 168 (Day 8) hours after dosing
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 2993.33 (280.33) | 3688.33 (525.56) | 4273.33 (947.49) | 2995.00 (568.99)

3. Primary Outcome: AUC0-inf
Description: Area under the curve (AUC0-inf) of ELX-02 plasma concentration following a single subcutaneous (SC) dose
Time Frame: 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24, 36, 48, 72, and 168 (Day 8) hours after dosing
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*ng/mL | 16997.41 (1776.84) | 35179.57 (9198.37) | 110925.53 (49098.37) | 15214.30 (2913.01)

4. Primary Outcome: Pharmacokinetic Parameters - Plasma Tmax
Description: Time to maximum concentration (Tmax) of ELX-02 plasma concentration following a single subcutaneous (SC) dose
Time Frame: 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, and 24 hours after dosing.
Measure: Median (Full Range); unit: hour
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour | 1.00 [0.75 to 2.00] | 1.00 [0.75 to 2.00] | 2.00 [1.00 to 6.00] | 1.50 [0.73 to 2.00]

5. Primary Outcome: Urine Pharmacokinetics Parameter - Ae0-t
Description: Cumulative amount of unchanged drug excreted into urine (Ae0-t) of ELX-02 following a single subcutaneous (SC) dose
Time Frame: Pre-dose (first void in the morning of Day 1), 0-3, 3-6, 6-9, 9-12, 12-18, 18-24, 24-36, 36-48, and 48-72 hours post-dose
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
mg | 61.50 (19.37) | 72.10 (26.45) | 54.86 (8.74) | 69.22 (17.70)

6. Primary Outcome: Urine Pharmacokinetic Parameter - Rmax
Description: Maximum rate of urinary extraction (Rmax) of ELX-02 following a single subcutaneous (SC) dose
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/h
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
mg/h | 9.18 (2.91) | 8.06 (5.91) | 3.11 (1.81) | 12.09 (2.82)

7. Primary Outcome: Number of Patients Reporting Treatment-Emergent Adverse Events (TEAEs) [Safety]
Description: TEAEs are undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the study treatment
Time Frame: 1-8 days
Measure: Number; unit: participants
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 0 | 0 | 2 | 9

ADVERSE EVENTS:
Time Frame: From the date of the signing of the consent form until follow-up visit on Day 8.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=6) | Group 2 (N=6) | Group 3 (N=6) | Group 4 (N=6)
Injection site erythema (General disorders) | 0 | 0 | 1 | 4
Injection site pruritus (General disorders) | 0 | 0 | 1 | 1
Injection site induration (General disorders) | 0 | 0 | 0 | 1
Blood pressure decrease (Investigations) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT03776539/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT03776539/SAP_001.pdf